CLINICAL TRIAL: NCT02290041
Title: Clinical Trial Phase I/II, of Test of Concept, Blind Double, Randomized, Controlled With Placebo, to Assess the Safety and Efficiency of the Treatment With Allogenic Adult Mesenchymal Stem Cells From Adipose Tissue Expanded, in HIV-infected Patients With Controlled Viremia and Immunological Discordant Response
Brief Title: Treatment With MSC in HIV-infected Patients With Controlled Viremia and Immunological Discordant Response
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Andalusian Initiative for Advanced Therapies - Fundación Pública Andaluza Progreso y Salud (Other)
Collaborators: Iniciativa Andaluza en Terapias Avanzadas (Other)
Responsible Party: Sponsor
Organization: Andalusian Network for Design and Translation of Advanced Therapies (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CeTMAd-VIH-2014
Record Dates: First submitted 2014-11-10; First posted 2014-11-13 (Estimated); Last update posted 2020-03-04 (Actual); Status verified 2020-03

CONDITIONS: Discordant Immunological Response in HIV Infected Subjects
Keywords: mesenchymal stem cells; HIV Infection; discordant immunological response
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Intervention Model Description: Phase 1: uncontrolled, single arm biosafety evaluation (n=5) Phase 2: placebo-controlled, randomized, evaluation (n=10)
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mesenchymal stem cells (Experimental): Intravenous infusion of 4 doses of allogenic adult mesenchymal stem cells from adipose tissue
  Interventions: Drug: Infusion of MSC
- Placebo (Placebo Comparator): Intravenous infusion of 4 doses of Placebo
  Interventions: Drug: Infusion of placebo

INTERVENTIONS:
Drug: Infusion of MSC — Intravenous infusion of 4 doses of adipose tissue derived allogeneic adult mesenchymal stem cells (1 million MSCs/Kg, weeks 0-4-8-20).
  Arms: Mesenchymal stem cells
Drug: Infusion of placebo — Infusion of placebo (weeks 0-4-8-20)
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
Phase I/IIClinical trial, proof of concept, double blind, and placebo-controlled, randomized 2:1 (MSCs: placebo), total sample size is 15 subjects

DETAILED DESCRIPTION:
This is a phase I-II, randomised, placebo-controlled, clinical trial, currently ongoing in a single Spanish hospital (Hospital Virgen del Rocío, Seville), to evaluate the safety and feasibility of a 4-doses treatment regimen with MSCs (1 million cells/Kg MSCs, weeks 0-4-8-20) in HIV infected adults with swith discordant virological and immunological response to antiretroviral therapy. In the initial phase of the trial (n=5), patients were sequentially recruited, with a safety period of 15 days, receiving unblinded cell therapy. In the second phase of the trial, subjects are block randomised (1:1) to receive either MSCs (n=5), or placebo (n=5), as the control treatment. Immune response variables, adverse events, opportunistic infection signs are evaluated as determinants of safety and efficacy of MSCs. Study endpoints are measured along a follow-up period of 24 months, that includes 17 visits according to a decreasing frequency rate. Intention to treat, and per protocol, and safety analysis will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed HIV infection
* Age> 18 years, both sexes
* In treatment with antiretroviral therapy (ART)
* Sustained HIV viral load <50 copies / ml for ≥ 1 years prior to study entry
* CD4 + cell count < 350/mL
* Immunological discordant response defined as: an increase <75 or <150 in CD4+ cell counts within one or two years of undetectable viraemia, respectively; or CD4 + cell count <350/mcl after 3 years of ART and undetectable viraemia (<50 copies/ml) ≥ 1 year
* Writen informed consent
* In women of child bearing potential or her partners:commitment to use contraceptive method of proved efficiency throughout the duration of the clinical trial

Exclusion Criteria:

* Pregnancy, breastfeeding, or refusal to the use of contraceptive methods
* Opportunistic infections in the last 12 months prior to study entry
* Active co-infection with hepatitis B virus/hepatitis C virus
* Child Pugh's scale stage C cirrhosis of the liver of any a aetiology
* Portal hypertension and / or hypersplenism of any aetiology
* Malignant neoplasia
* Treatment with steroids, immunomodulators, interferon, chemotherapy or any other medicinal product that could modify the number of CD4+ within the last 12 months prior to study entry
* Confirmed analytical 3 or 4 grade (AIDS Clinical Trials Group scale) abnormalities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2017-02-08 (Actual); Primary Completion 2019-07-30 (Actual); Study Completion 2019-07-30 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse reactions | 24 months
  Incidence of adverse reactions grade 3 and 4 according to DAIDs scale
Incidence of opportunist diseases | 24 months
Changes in CD4+ cell count and CD4+/CD8+ ratio | 28 days after the 4th infusion MSCs/placebo
  Changes in CD4+ cell count and CD4+/CD8+ ratio as measured by flow citometry

SECONDARY OUTCOMES:
T CD4 +/µl count evolution and CD4 +/CD8 + ratio throughout 48 weeks | 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Luis F. López Cortés, MD, Study Chair — Hospitales Universitarios Virgen del Rocío
Locations (1):
- Virgen del Rocío University Hospital, Seville, Spain

REFERENCES:
- [Derived] Trujillo-Rodriguez M, Viciana P, Rivas-Jeremias I, Alvarez-Rios AI, Ruiz-Garcia A, Espinosa-Ibanez O, Arias-Santiago S, Martinez-Atienza J, Mata R, Fernandez-Lopez O, Ruiz-Mateos E, Gutierrez-Valencia A, Lopez-Cortes LF. Mesenchymal stromal cells in human immunodeficiency virus-infected patients with discordant immune response: Early results of a phase I/II clinical trial. Stem Cells Transl Med. 2021 Apr;10(4):534-541. doi: 10.1002/sctm.20-0213. Epub 2020 Dec 2. PMID 33264515